CLINICAL TRIAL: NCT05462080
Title: Correlation of Motor Metrics and Neurological Data (COMMAND)
Brief Title: Correlation of Motor Metrics and Neurological Data
Acronym: COMMAND
Status: Completed | Type: Observational
Sponsor: Ceraxis Health, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: REDD 0001
Record Dates: First submitted 2022-07-06; First posted 2022-07-18 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Movement Disorders (Incl Parkinsonism)
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Movement Disorders Patients
  Interventions: Diagnostic Test: Ceraxis product

INTERVENTIONS:
Diagnostic Test: Ceraxis product — All patients will have their symptoms evaluated using the Ceraxis product

SUMMARY:
This is a pilot study to collect data with the Ceraxis product and standard movement disorders tests in order to prove and codify potential correlations.

ELIGIBILITY:
Inclusion Criteria:

* Adult with a diagnosis of idiopathic Parkinson's disease or essential tremor by a movement disorders neurologist
* Age greater than or equal to 21 years
* Hoehn and Yahr stage I-III
* Ability to ambulate 200+ meters independently
* Ability to follow 2-step commands
* Clinically responsive to medication or Deep Brain Stimulation (DBS)
* Clinically optimized medication or DBS for at least six months
* Able to tolerate withdrawal of medication and/or DBS

Exclusion Criteria:

* Any comorbidity which would exclude them from being able to use the Ceraxis product
* Inability to learn how to use the system
* Diagnosis of dementia or impairment that compromises the ability to provide informed consent
* Neurological disease other than Parkinson's disease or essential tremor (i.e. multiple sclerosis, stroke with residual motor deficits)
* Musculoskeletal injury that significantly alters gait

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Movement disorders patients being treated at the site
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Collection of data with Ceraxis product (stylus product with a built-in Inertial Measurement Unit (IMU) which includes a 3-axis accelerometer, gyroscope, and magnetometer, as well as a force sensing tip) | Day 1
  Patients will be guided through a set of actions while the sensors record movement data on their upper and lower extremity motor symptoms. This data will be correlated with the secondary outcome measures post hoc.

SECONDARY OUTCOMES:
UPDRS-I, UPDRS-II, and UPDRS-III assessment for patients with Parkinson's disease | Day 1
TETRAS tremor rating scale for patients with Essential Tremor | Day 1
Upper extremities motor strength, assessed by neurological examination | Day 1
Coordination test for the upper extremities to evaluate dysdiadochokinesia | Day 1
Archimedes Spiral task | Day 1
Freezing of Gait questionnaire | Day 1
Usage Survey | Day 1
  Custom survey given to patients to collect their impressions of the Ceraxis product

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided